CLINICAL TRIAL: NCT01435096
Title: A Phase I Dose Finding Study of BN80927 Administered as an Intravenous Infusion Once Every 3 Weeks in Patients With Advanced Malignant Solid Tumors
Brief Title: BN80927 in Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-55-52905-701; 2005-002703-16 (EudraCT Number)
Record Dates: First submitted 2011-08-24; First posted 2011-09-15 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Malignant Solid Tumour
MeSH Terms: interventions — BN 80927

ARMS (1):
- BN80927 (Experimental)
  Interventions: Drug: BN80927

INTERVENTIONS:
Drug: BN80927 — Administered over 30 minutes in the vein with a fixed infusion rate once every 3 weeks. Each patient could participate in a maximum of 10 continuous cycles, equivalent to 30 weeks treatment.

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose and the recommended dose of BN80927 in patients with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

All included patients:

* Gave their written (personally signed and dated) informed consent
* had histologically or cytologically documented malignant solid tumour
* had received no more than three prior chemotherapy regimens
* had failed the standard therapy or had no option of an active standard therapy
* had an estimated survival time of greater than 3 months (according to the investigator's assessment)
* had a World Health Organisation (WHO) performance status score ≤1
* were free from other serious concurrent disease
* had adequate bone marrow function
* had adequate liver function
* had adequate renal function
* who were female and of child-bearing potential must have had a negative result in a pre-study pregnancy test β-human-chorionic-gonadotrophin (β-HCG).

Exclusion Criteria:

No patient included:

* was pregnant or lactating
* was unable and/or unwilling to comply fully with the protocol and the study instructions;
* presented with any concomitant condition, which could compromise the objectives of the study
* had received an investigational drug within 30 days prior to study entry or was scheduled to require concurrent treatment with an experimental drug or treatment during the study
* had received chemotherapy or hormonotherapy within 4 weeks of study entry, or had received chemotherapy with nitrosoureas or mitomycin-C within 6 weeks of study entry
* had received any extensive palliative or curative radiotherapy (no more than 35% of their active bone marrow) within 2 weeks of study entry, or had not fully recovered from such treatment
* had previously received a bone marrow transplant (BMT) or peripheral blood progenitor cells (PBPC)
* had clinical evidence of major organ failure or brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by incidence of dose limiting toxicity. | During cycle 1, up to 3 weeks
Recommended dose determined by incidence of dose limiting toxicity. | During cycle 1, up to 3 weeks

SECONDARY OUTCOMES:
Tumour response assessment according to the Response Evaluation Criteria in Solid Tumours (RECIST) criteria. | Baseline, week 3 of cycle 2, then on alternate cycles of treatment (maximum 10 cycles, up to 30 weeks)
Cmax | 72 hours post-dose in treatment cycle 1 and 2 (each cycle is 21 days)
Area Under Curve | 72 hours post-dose in treatment cycle 1 and 2 (each cycle is 21 days)
Tmax | 72 hours post-dose in treatment cycle 1 and 2 (each cycle is 21 days)
T1/2 | 72 hours post-dose in treatment cycle 1 and 2 (each cycle is 21 days)
Number of adverse events | Monitored weekly at all treatment cycles and the end of study visit. Maximum 10 treatment cycles, up to 30 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (3):
- France (3):
  - Centre Paul Papin, Angers
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud